CLINICAL TRIAL: NCT01938157
Title: Diffusion Weighted MR Imaging of the Breasts in Women at High Risk of Breast Cancer: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12-2327
Record Dates: First submitted 2013-08-19; First posted 2013-09-10 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: High Risk of Breast Cancer; Diffusion Magnetic Resonance Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Risk Breast Cancer Patients (Experimental): High Risk Breast Cancer Patients (all subjects)
  Interventions: Procedure: Diffusion-weighted MR imaging

INTERVENTIONS:
Procedure: Diffusion-weighted MR imaging — An addition 90 seconds of DWI will be added to a clinical breast MRI for all patients agreeing to participate in the study.

SUMMARY:
Purpose: The purpose of this pilot study is to evaluate whether MRI of the breasts with diffusion-weighted MR imaging can identify features more specific for breast cancer in women at high-risk of developing breast cancer.

Participants: One hundred asymptomatic women at high-risk for breast cancer recommended for a clinical breast MRI identified through the UNC Breast Clinic will be consecutively recruited for this study.

Procedures (methods): Each patient will undergo a clinical breast MRI and the addition of a single 90 second diffusion weighted sequence. A reader study will be conducted at UNC after the completion of patient accrual. The images will be analysed for lesions, enhancement patterns, diffusion weighted imaging data and correlated with any pathology or 1 year follow-up MRI exam. The study information will be entered into a secure database and analyzed.

DETAILED DESCRIPTION:
Enrollment and Recruitment:

A total of 100 high-risk women will be enrolled in this pilot study. High-risk for this study is defined as women at significantly increased risk of breast cancer. The Investigators will use the American Cancer Society Guidelines for Breast Screening with MRI as adjunct to mammography [2]. These guidelines recommend annual screening mammography for high risk women including BRCA mutations, first-degree relative of BRCA carrier, lifetime risk 20-25% or greater, previous history of chest radiation age 10 to 30 years and other syndromes related to increased breast cancer risk. We also included women with a history of previous high risk breast lesion(s) such as atypical hyperplasia, lobular carcinoma in situ or atypical lobular hyperplasia and a personal history of breast cancer by clinical consensus.

Patients who have been scheduled for the study will be contacted by research staff by phone to ask if they would be interested in participating in a research study. A script will be used to determine if patient is interested in hearing about a research study, if not the call will be discontinued immediately. If yes, more details will be provided to the patient to make a determination if they would like to participate.

If the patient is interested, she will be asked to come into the UNC MRI Department one hour prior to her scheduled MRI appointment. On the day of her MRI study, the patient will meet with the study coordinator or other assigned listed study personnel and will consent the subject to this study. Research coordinator/listed study personal will go through the consent form with the patient and answer any questions she may have. If patient agrees to participate after review of consent form, the patient will sign and date, the coordinator will then sign and date and patient will be formally enrolled. The patient will then undergo her ordered clinical breast MRI followed by one diffusion weighted MRI sequence.

Imaging Procedure: Each eligible patient, who provides consent for the study, will undergo a MR imaging screening questionnaire. If the patient has no contraindications, an intravenous line will be placed into a vein in the patient's arm and the patient will be placed prone with her breasts in a dedicated MRI breast coil. The patient will be given earplugs to decrease the noise level while in the magnet during the 45 minute total time period. High-resolution MRI sequences of the breasts and axillary regions will be performed before and after a gadolinium-DTPA bolus injection as per ordered clinical breast MRI protocol. Afterwards, one diffusion-weighted (DW) MRI sequence of the breast(s) will be performed. The DW sequence takes approximately 90 seconds.

The clinical images will be interpreted as per clinical protocol. The clinical radiologists will not have DW images to interpret. Therefore, it will not influence clinical decision concerning therapy.

Needle Core Biopsy/Surgery: All patients who are recommended for a needle core biopsy or open surgical biopsy for a breast lesion from their clinical Breast MRI will be scheduled by their surgeon. The radiologist performing the MRI-guided needle core biopsy or the surgeon performing the open surgical biopsy will be blinded to the results of the DW imaging, and therefore it will not influence clinical decision concerning therapy.

Reader Study: Five readers, radiologists that are experts in breast imaging and who are blinded to the study results, will be given de-identified MRI and DWI MRI images from the patient's entry MRI (MRIe) study and 1-year follow-up MRI (MRIf) study. Study radiologist data sheets will be completed for each study. The reader will have to complete the data sheets for MRIe before he/she can read and evaluate MRIf. The readers are blinded to the pathologic data at all times. For each condition MRIe and MRIf, each reader will check one of the checkboxes of each query that presents the lesion type (mass or non-mass enhancement), anatomic location (upper outer, upper inner, lower outer, lower inner or subareolar), largest dimension in centimeter, signal intensity on T1- and T2-weighted images (high, iso- or low to the fibroglandular tissue), morphology such as shape (round, oval, lobulated or irregular) and margin(smooth, irregular or spiculated) for mass, distribution (focal, linear, ductal, segmental or regional) for non-mass enhancement, enhancement pattern (homogeneous, heterogeneous, rim enhancement, dark internal septations, enhancing internal septations or central enhancement for mass; homogeneous, heterogeneous, stippled/punctate, clumped or reticular/dendritic for non-mass enhancement) and kinetic curve patterns on contrast-enhanced MRI (persistent, plateau or washout), signal intensity on DWI MRI /ADC map (high, iso-, low to the fibroglandular tissue) and an ADC value marked through quantitative analysis on the DWI study. The readers will assign any lesion(s) as benign, probably benign, suspicious and highly suggestive of malignancy according to the imaging findings and decide the probability of malignancy in percentages on contrast-enhanced MRI and DWI MRI, independently for the entry and final MRI study. After each radiologist reader has completed the data sheets for each patient, the data will be entered into a secure data base for statistical analysis.

ELIGIBILITY:
Inclusion Criteria

1. Women at high-risk of breast cancer with an order for a clinical screening breast MRI.
2. Asymptomatic women.
3. Able to provide informed consent.
4. At least 21 years of age.

Exclusion Criteria

1. Women with symptom such as palpable mass or nipple discharge.
2. Women with MRI/MRA contraindications such as a cardiac pacemaker, and aneurysm clip, cochlear implants, and metal in the eyes.
3. Women who have had a moderate or severe contrast reaction to intravenous gadolinium-DTPA.
4. Women who are not able to give consent.
5. Women diagnosed with breast cancer within the last 6 months.
6. Women who are pregnant.
7. Male patients.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Number of identified lesions | 1 year from screening imaging
  Lesions will be identified by 5 trained radiologists in a reader study. The identification of lesions will be confirmed by pathologists, or if no biopsy is performed, then truth will be determined after a 1-year follow-up MRI/MRI DWI.

SECONDARY OUTCOMES:
A composite of the sensitivity, specificity, and AUC of contrast-enhanced MRI and diffusion MRI | 1 year following screening imaging
  Trained radiologists will complete a series of questionnaires about identified lesions. Using these questionnaires, a mixed-effect ANOVA model (Obuchowski and Rockette, 1995) is to fit these summary measures of diagnostics accuracy. To test the primary hypothesis , an approximately t-distributed statistic based on Obuchowski and Rockette (1995) will be used and we reject the hypothesis if the statistic is larger than 95% percentile of a central student's t-distribution with one degree of freedom.

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Kuzmiak, DO, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States